CLINICAL TRIAL: NCT07212439
Title: Continuous Cough Monitoring for Early Detection of COPD Exacerbations Using Hyfe
Brief Title: Monitoring Coughs for the Early Detection of Worsening COPD
Acronym: Hyfe-EPOC
Status: Recruiting | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Hyfe Inc (Other)
Responsible Party: Sponsor
Other Study IDs: Hyfe-EPOC
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; COPD Exacerbation; Cough; Cough Monitoring; Hyfe; Early Detection; Wearable Device; Artificial Intelligence; Observational Study
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inpatients: This cohort consists of patients with a confirmed COPD diagnosis who are currently hospitalized due to a severe COPD exacerbation.
- Outpatients: This cohort includes outpatients with a COPD diagnosis who are being seen for routine follow-up. To be included, these patients must have a history of at least one exacerbation in the past 12 months.

SUMMARY:
This study is for adults with COPD. Flare-ups of COPD, also known as exacerbations, can be serious and lead to hospital stays. The purpose of this research is to see if continuously and automatically monitoring a person's coughs can help predict these flare-ups early, before they become severe. Participants will use the Hyfe cough monitoring system, which includes a watch-like device worn on the wrist and a smartphone application. The system privately counts the number of coughs without recording any audio. Participants will also answer a short, weekly questionnaire about their COPD symptoms. This is an observational study, which means it will not change the regular medical care a participant receives. The participants and their care providers will not see the cough counts. The doctor will continue to manage their COPD as usual.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational cohort study designed to evaluate the accuracy of a continuous, passive acoustic monitoring system (Hyfe) for the early detection of COPD exacerbations. COPD exacerbations are a major driver of disease progression and healthcare utilization, but current detection methods rely on subjective patient-reported symptoms. Cough is a core symptom of COPD, and its objective quantification may provide an early warning signal for clinical worsening. This study aims to determine if changes in cough frequency, as measured by the Hyfe system, can predict an upcoming exacerbation with a clinically relevant lead time. The study will enroll two cohorts of patients with a COPD diagnosis: outpatients with a history of frequent exacerbations and inpatients hospitalized for a severe exacerbation. Participants will use the Hyfe Cough Monitor Suite to continuously track cough frequency and will complete the COPD Assessment Test (CAT) questionnaire weekly. To ensure an unbiased assessment, treating clinicians will be blinded to all study-collected data (both cough counts and CAT scores). The clinical diagnosis of a COPD exacerbation, as defined by GOLD 2025 criteria and made by the blinded clinician, will serve as the ground truth endpoint.

ELIGIBILITY:
Inclusion criteria:

* Must be 18 years of age or older.
* Must have an existing diagnosis of COPD.
* For the inpatient cohort, participants must be currently assessed as having a moderate/severe exacerbation.
* For the outpatient cohort, participants must have had at least one exacerbation of any severity in the last 12 months.
* For the outpatient cohort, at least one month must have passed since the last exacerbation.

Exclusion criteria:

* Individuals who are unable to provide informed consent.
* Individuals who are unable to adhere to study procedures.
* For the inpatient cohort, individuals requiring invasive or non-invasive ventilation.
* Individuals who live with a person who has a chronic cough.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll adult participants with a confirmed diagnosis of COPD. The population is composed of two distinct groups: inpatients who are currently hospitalized for a moderate/severe COPD exacerbation, and outpatients attending routine follow-up who are selected to enrich the sample with individuals who experience frequent exacerbations.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Predictive accuracy of Hyfe cough monitoring for COPD exacerbations | Up to 1 year
  (a) Positive predictive value (PPV) by time to exacerbation vs standard of care (SoC) (b) False positive and false negative rates by time to exacerbation vs SoC

SECONDARY OUTCOMES:
Predictive accuracy: continuous vs. nighttime-only cough monitoring | Up to 1 year
  Positive predictive value by time to exacerbation of continuous vs night-only monitoring
Predictive accuracy: cough data vs. combined cough and symptom data | Up to 1 year
  Positive predictive value by time to exacerbation of cough monitoring with and without the COPD Assessment Test (CAT) questionnaire vs the standard of care
Estimated potential cost savings | Up to 1 year
  Derived from hospitalization rate and 30-day readmission rates from standard of care vs the expected rates with earlier detection through cough monitoring should there be any
Usability and acceptability of the Hyfe monitoring system | Up to 1 year
  Usability will be measured by participant adherence, calculated as the percentage of time the monitor is worn or actively charging. Acceptability will be assessed using a self-reported user satisfaction survey administered to participants at the end of their follow-up period

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Clinica San Miguel, Pamplona, Navarre
  - Clínica Universidad de Navarra, Universidad de Navarra, Pamplona, Navarre
  - Servicio Navarro de Salud, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: No
The study protocol does not outline a plan for sharing IPD with researchers external to the study team. The protocol's dissemination plan is focused on sharing aggregated study results in scientific meetings and through publication in peer-reviewed journals. While anonymized data will be shared with the study's co-investigators and the sponsor, there is no provision for making IPD available to other researchers.

REFERENCES:
- [Background] Mackay AJ, Donaldson GC, Patel AR, Jones PW, Hurst JR, Wedzicha JA. Usefulness of the Chronic Obstructive Pulmonary Disease Assessment Test to evaluate severity of COPD exacerbations. Am J Respir Crit Care Med. 2012 Jun 1;185(11):1218-24. doi: 10.1164/rccm.201110-1843OC. Epub 2012 Jan 26. PMID 22281834
- [Background] Folch Ayora A, Macia-Soler L, Orts-Cortes MI, Hernandez C, Seijas-Babot N. Comparative analysis of the psychometric parameters of two quality-of-life questionnaires, the SGRQ and CAT, in the assessment of patients with COPD exacerbations during hospitalization: A multicenter study. Chron Respir Dis. 2018 Nov;15(4):374-383. doi: 10.1177/1479972318761645. Epub 2018 Mar 12. PMID 29529879
- [Background] Jones PW, Brusselle G, Dal Negro RW, Ferrer M, Kardos P, Levy ML, Perez T, Soler Cataluna JJ, van der Molen T, Adamek L, Banik N. Properties of the COPD assessment test in a cross-sectional European study. Eur Respir J. 2011 Jul;38(1):29-35. doi: 10.1183/09031936.00177210. Epub 2011 May 12. PMID 21565915
- [Background] Kim V, Aaron SD. What is a COPD exacerbation? Current definitions, pitfalls, challenges and opportunities for improvement. Eur Respir J. 2018 Nov 15;52(5):1801261. doi: 10.1183/13993003.01261-2018. Print 2018 Nov. PMID 30237306
- [Background] Gabaldon-Figueira JC, Keen E, Rudd M, Orrilo V, Blavia I, Chaccour J, Galvosas M, Small P, Grandjean Lapierre S, Chaccour C. Longitudinal passive cough monitoring and its implications for detecting changes in clinical status. ERJ Open Res. 2022 May 16;8(2):00001-2022. doi: 10.1183/23120541.00001-2022. eCollection 2022 Apr. PMID 35586452
- [Background] Gabaldon-Figueira JC, Keen E, Gimenez G, Orrillo V, Blavia I, Dore DH, Armendariz N, Chaccour J, Fernandez-Montero A, Bartolome J, Umashankar N, Small P, Grandjean Lapierre S, Chaccour C. Acoustic surveillance of cough for detecting respiratory disease using artificial intelligence. ERJ Open Res. 2022 May 30;8(2):00053-2022. doi: 10.1183/23120541.00053-2022. eCollection 2022 Apr. PMID 35651361
- [Background] Chung KF, Chaccour C, Jover L, Galvosas M, Song WJ, Rudd M, Small P. Longitudinal Cough Frequency Monitoring in Persistent Coughers: Daily Variability and Predictability. Lung. 2024 Oct;202(5):561-568. doi: 10.1007/s00408-024-00734-x. Epub 2024 Jul 31. PMID 39085518
- [Background] Chaccour C, Sanchez-Olivieri I, Siegel S, Megson G, Winthrop KL, Botella JB, de-Torres JP, Jover L, Brew J, Kafentzis G, Galvosas M, Rudd M, Small P. Validation and accuracy of the Hyfe cough monitoring system: a multicenter clinical study. Sci Rep. 2025 Jan 6;15(1):880. doi: 10.1038/s41598-025-85341-3. PMID 39762316
- [Background] den Brinker AC, Thackray-Nocera S, Crooks MG, Morice AH. Improved Precision of COPD Exacerbation Detection in Night-Time Cough Monitoring. J Pers Med. 2025 Aug 2;15(8):349. doi: 10.3390/jpm15080349. PMID 40863411
- [Background] Morice AH, den Brinker AC, Crooks M, Thackray-Nocera S, Ouweltjes O, Rietman R. Can Passive Cough Monitoring Predict COPD Exacerbations? COPD. 2025 Apr 4;22(1):2487909. doi: 10.1080/15412555.2025.2487909. Epub 2025 Apr 14. PMID 40223505